CLINICAL TRIAL: NCT00588133
Title: A Preliminary Study of a New Tranexamic Acid Dosing Schedule for Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Gregory A. Nuttall, M.D., Mayo Clinic College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1216-00
Record Dates: First submitted 2007-12-25; First posted 2008-01-08 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Cardiac Surgery
Keywords: antifibrinolytic, bleeding, heart
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): New drug dosing schedule
  Interventions: Drug: tranexamic acid
- 2 (Active Comparator): Standard drug dosing schedule
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — Loading dose: 6.6 mg/kg Prime dose: 50 mg for 2.5 Liter circuit (assuming 1 L/kg Vd in prime fluids), 40 mg for 2 Liter circuit Rate of infusion: 6 mg/kg/hr
  Renal Insufficiency (normal loading dose and prime dose):
  Serum Creatinine = 1.6-3.3: reduce infusion to 4.5 mg/kg/hr Serum Creatinine = 3.3-6.6: reduce infusion to 3.0 mg/kg/hr Serum Creatinine = >6.6: reduce infusion to 1.5 mg/kg/hr
  Other Names: Cyclokapron
  Arms: 1
Drug: tranexamic acid — 10 mg/kg tranexamic acid given over 20 minutes followed by an infusion of 1 mg/kg/hr
  Other Names: Cyclokapron
  Arms: 2

SUMMARY:
Tranexamic acid is administered intravenously to prevent bleeding associated with cardiac surgery and cardiopulmonary bypass. We have developed an assay for tranexamic acid. We have developed an alternative dosing schedule for tranexamic acid. The objective of this preliminary study is to determine if this new dosing schedule can achieve the desired plasma concentration of tranexamic acid and reduce intra and inter patient variability in tranexamic acid plasma concentrations relative to the current dosing schedule.

DETAILED DESCRIPTION:
Tranexamic acid is administered intravenously to prevent bleeding associated with cardiac surgery and cardiopulmonary bypass. The current dosing regimen for tranexamic acid was empirically derived based upon pharmacokinetics in normal patients receiving the drug. We have developed an assay for tranexamic acid and found that the plasma concentration of tranexamic acid varies greatly between patients and also over time within each patient, especially in patients with renal insufficiency. We have developed an alternative dosing schedule for tranexamic acid that incorporates the effects of renal function on tranexamic acid concentrations. The objective of this preliminary study is to determine if this new dosing schedule can achieve the desired plasma concentration of tranexamic acid and reduce intra and inter patient variability in tranexamic acid plasma concentrations relative to the current dosing schedule. The results of this study will be used in a larger subsequent study of what level of plasma tranexamic acid concentration is needed to prevent bleeding and transfusion of blood products in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or greater having cardiac surgery.

Exclusion Criteria:

* Age less than 18 years old.
* Since tranexamic acid is not approved for pregnant patients, those extremely rare patients that are pregnant and having cardiac surgery will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Plasma tranexamic acid levels | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Nuttall, M.D., Principal Investigator — Mayo Clinic College of Medicine